CLINICAL TRIAL: NCT01135264
Title: Gambling Addiction: Treatment Mediators and Moderators
Brief Title: Cognitive-Motivational Behavior Therapy for Pathological Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #5946/6970R; 1R01MH082773-01A1 (NIH); 1R01MH082733-01A1 (NIH)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-01

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Active Comparator): The CBT treatment developed by Ladouceur (Consultant) will serve as control condition (outline of published treatment manual by Ladouceur & Lachance, 2006. This treatment served as a model for the cognitive-behavioral component in CMBT and has received empirical support in two studies from Ladouceur's lab (Sylvain et al., 1997; Ladouceur et al., 2004). It places strong emphasis on cognitive correction of erroneous beliefs about gambling and also focuses on coping skills training and relapse prevention. CBT also lasts 12 weekly sessions.
  Interventions: Behavioral: CBT
- CMBT (Experimental): We used the NIMH-funded R21 mechanism to develop and test the CMBT intervention (Wulfert et al., 2003, 2005; 2006). Treatment will be implemented in 12 weekly sessions (3 motivational enhancement sessions, 8 sessions of cognitive-behavioral treatment, 1 session of relapse prevention)
  Interventions: Behavioral: CMBT

INTERVENTIONS:
Behavioral: CBT — The CBT treatment developed by Ladouceur (Consultant) will serve as control condition (outline of published treatment manual by Ladouceur & Lachance, 2006. This treatment served as a model for the cognitive-behavioral component in CMBT and has received empirical support in two studies from Ladouceur's lab (Sylvain et al., 1997; Ladouceur et al., 2004). It places strong emphasis on cognitive correction of erroneous beliefs about gambling and also focuses on coping skills training and relapse prevention. CBT also lasts 12 weekly sessions.
  Arms: CBT
Behavioral: CMBT — We used the NIMH-funded R21 mechanism to develop and test the CMBT intervention (Wulfert et al., 2003, 2005; 2006). Treatment will be implemented in 12 weekly sessions (3 motivational enhancement sessions, 8 sessions of cognitive-behavioral treatment, 1 session of relapse prevention)
  Arms: CMBT

SUMMARY:
In the proposed two-arm randomized controlled trial, 200 patients meeting DSM-IV criteria for PG will be randomized to 12 sessions of Cognitive-Motivational Behavior Therapy (CMBT) or to Cognitive Behavior Therapy (CBT).

DETAILED DESCRIPTION:
CMBT has been developed by our team over the last five years, and has shown very promising results in a small, NIMH-funded randomized pilot trial (R21 MH 064568). We will assess patients biweekly during the active treatment phase and follow them for 12 months after the end of treatment to obtain data on long-term treatment outcome. We hypothesize that CMBT will show higher efficacy and retention than CBT in the treatment phase, and that gains will be maintained at a higher rate during follow-up.

A second major purpose of the proposed study is to elucidate the presumed mechanisms of change by examining potential mediators (readiness to change, irrational beliefs about gambling, coping skills, therapeutic alliance) and moderators (psychiatric comorbidity with Axis I and II disorders, family history of PG, impulsivity, and baseline motivation to change) of treatment response. A better understanding of how the proposed interventions work will help advance the science and treatment of PG and will be helpful in the future refinement and adaptation of CMBT. Identifying patient subgroups for which the intervention is particularly effective is essential for rational treatment selection. Thus, the immediate goal of the project is to compare CBMT versus CBT for the treatment of PG. A long-term goal of the proposed research is to establish effective treatment procedures that reduce the considerable individual and social costs of PG.

ELIGIBILITY:
Inclusion Criteria:

* pathological gambling
* be able to read, understand and sign an informed consent form prior to any procedure and must be willing to comply with all study procedures and timelines

Exclusion Criteria:

* to meet DSM-IV criteria for comorbid substance use disorders in the last six months
* current comorbid psychiatric conditions which require treatment and are not clearly secondary to pathological gambling
* psychotropic medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
patient retention | 60 weeks
  Retention will be measured by the number of treatment sessions attended

SECONDARY OUTCOMES:
gambling behavior | 60 weeks
  Our primary measure will be money lost gambling. Secondary measures will include days gambled; scores on the PG-YBOCS, proportion of patients meeting diagnosis of PG and of those having achieved abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Blanco, M.D., Principal Investigator — New York Psychiatric Institute
Locations (1):
- New York Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Blanco C, Potenza MN, Kim SW, Ibanez A, Zaninelli R, Saiz-Ruiz J, Grant JE. A pilot study of impulsivity and compulsivity in pathological gambling. Psychiatry Res. 2009 May 15;167(1-2):161-8. doi: 10.1016/j.psychres.2008.04.023. Epub 2009 Apr 1. PMID 19339053
- [Background] Blanco C, Hasin DS, Petry N, Stinson FS, Grant BF. Sex differences in subclinical and DSM-IV pathological gambling: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Psychol Med. 2006 Jul;36(7):943-53. doi: 10.1017/S0033291706007410. Epub 2006 May 2. PMID 16650342
- [Background] Okuda M, Balan I, Petry NM, Oquendo M, Blanco C. Cognitive-behavioral therapy for pathological gambling: cultural considerations. Am J Psychiatry. 2009 Dec;166(12):1325-30. doi: 10.1176/appi.ajp.2009.08081235. PMID 19952084
- [Background] Wulfert E, Blanchard EB, Freidenberg BM, Martell RS. Retaining pathological gamblers in cognitive behavior therapy through motivational enhancement: A pilot study. Behav Modif. 2006 May;30(3):315-40. doi: 10.1177/0145445503262578. PMID 16574817
- [Background] Wulfert E, Maxson J, Jardin B. Cue-specific reactivity in experienced gamblers. Psychol Addict Behav. 2009 Dec;23(4):731-5. doi: 10.1037/a0017134. PMID 20025381
- [Background] Wulfert E, Franco C, Williams K, Roland B, Maxson JH. The role of money in the excitement of gambling. Psychol Addict Behav. 2008 Sep;22(3):380-390. doi: 10.1037/0893-164X.22.3.380. PMID 18778131